CLINICAL TRIAL: NCT02080910
Title: The Effects of a Psychoeducational Intervention on Stroke Family Caregiver Outcomes and the Use of Health and Social Services Among Stroke Survivors: A Randomized Controlled Trial
Brief Title: A Psychoeducational Intervention for Stroke Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ho Yu CHENG, PhD (Nursing) candidate, BN, PgD (Mental Health), RN, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CRE-2012.185-T
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Stroke
Keywords: Caregiver; stroke; psychoeducation; problem-solving
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychoeducational program (Experimental): Psychoeducational program consisted of (1) two inpatient sessions of face-to-face education on stroke and its caregiving; (2) six biweekly problem-solving training via telephone contacts after the discharge of stroke survivors
  Interventions: Behavioral: Psychoeducation
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Psychoeducation
  Arms: Psychoeducational program

SUMMARY:
This is a randomized controlled trial with a 3-month psychoeducational program as intervention, followed by a 3 month observational period. The purpose of this study was to examine whether a psychoeducational program focusing on equipping caregivers with problem-solving skills would improve caregiver's problem-solving abilities, their psychological responses and caregiving resources, and would minimize the use of health and social services among stroke survivors.

ELIGIBILITY:
Inclusion Criteria (caregiver):

* Family member of stroke survivor
* Chinese adult
* Live with stroke survivors
* Primary caregiver
* Being able to communicate with the researcher

Inclusion Criteria (stroke survivor):

* Chinese adult with diagnosis of stroke
* Live at home after discharge
* Being able to understand and to give consent

Exclusion Criteria (caregiver and stroke survivor):

* History of self-reported doctor-diagnosed psychiatric illness
* (stroke survivor): being mild to totally independent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Caregivers' change in depressive symptom severity from baseline | 3 month post intervention
  Change in depressive symptoms severity, as measured by the 10-item Center for Epidemiological Studies Depression (Chinese version), will be analyzed by the GEE model
Caregiver's change in perceived mental health from baseline | 3 months post intervention
  Change in perceived mental health, as measured by the Chinese (Hong Kong) Medical Outcomes Study 12-item Short Form Health Survey version 2 (SF-12v2), its mental component summary score will be analyzed by the GEE model
Caregiver's change in caregiving burden | at immediate post-intervention, 1-month post-intervention, 3-month post-intervention
  End-point between-group differences of the caregiving burden, as measured by the Caregiving Strain Index (Chinese version), will be analyzed by multiple regression analysis
Caregiver's change in caregiving competence from baseline | 3 months post intervention
  Change in caregiving competence, as measured by the Caregiving Competence Scale (Chinese version), will be analyzed by the GEE model

SECONDARY OUTCOMES:
Caregiver's change in self-appraised problem-solving abilities from baseline | 3 months post intervention
  Change in self-appraised problem-solving abilities, as measured by the Problem Solving Inventory (Chinese version), will be analyzed using the Generalized Estimating Equations (GEE) model
Caregiver's change in family functioning from baseline | 3 months post intervention
  Change in family functioning, as measured by the McMaster Model of Family Assessment Device (Chinese version), will be analyzed using the GEE model
Caregiver's change in perceived social support from baseline | 3 months post intervention
  Change in perceived social support, as measured by the Six-item Social Support Questionnaire (Chinese version), will be analyzed using the GEE model
Caregiver's change in perceived physical health from baseline | 3 months post intervention
  Change in perceived physical health, as measured by the Chinese (Hong Kong) SF-12v2 (Physical Component Summary Score), will be analyzed by the GEE model
Caregiving-related injuries | at immediate post-intervention, 1-month post-intervention, 3-month post-intervention
  End-point between-group differences of the self-reported caregiving related injuries will be analyzed using Chi square statistics
Stroke-related hospital readmission (stroke survivors) | at immediate post-intervention, 1-month post-intervention, 3-month post-intervention
  End-point between-group differences of the self-reported stroke-related hospital readmission, such as falls, recurrent stroke, will be analyzed using Chi square statistics
Placement to residential/nursing care home (stroke survivors) | at immediate post-intervention, 1-month post-intervention, 3-month post-intervention
  End-point between-group differences of the placement to residential/nursing care home of stroke survivors will be analyzed by the Chi square statistics

CONTACTS AND LOCATIONS:
Overall Officials: Ho Yu CHENG, PgD (MH), BN, Principal Investigator — Nethersole School of Nursing, Chinese University of Hong Kong; Janita Chau, PhD, Study Chair — The Nethersole School of Nursing
Locations (1):
- Prince of Wales Hospital, Shatin Hospital, Tai Po Hospital, Hong Kong SAR, China

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082